CLINICAL TRIAL: NCT06992921
Title: Towards Personalized Nutrition With SCAPIS2-HOME - Dissecting Determinants of Interpersonal Metabolic Responses to Standardized Meals and Mixed Meal Tolerance Tests
Brief Title: Towards Personalized Nutrition With SCAPIS2-HOME
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chalmers University of Technology (Other)
Collaborators: Göteborg University (Other); Umeå University (Other); Hjärt-Lungfonden, Sweden (Unknown); Lantmännen (Unknown)
Responsible Party: Principal Investigator, Rikard Landberg, Professor, Chalmers University of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SCAPIS2-HOME
Record Dates: First submitted 2025-04-30; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Disease (CVD); Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Personalized nutrition; Precision nutrition; Mixed meal tolerance test; Continuous glucose monitoring; Home sampling
MeSH Terms: conditions — Cardiovascular Diseases; Pulmonary Disease, Chronic Obstructive | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dietary intervention (Experimental): 10-day dietary intervention using standardized test meals
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — Iterventional dietary study using standardised meals with different fat content and carbohydrate quantity and quality or mixed meal tolerance test to predict for an individuals metabolic response.

SUMMARY:
The Swedish CardioPulmonary bioImage Study (SCAPIS) is a nationwide, open-access, population-based cohort in Sweden designed to study cardiovascular disease and chronic obstructive pulmonary disease. In January 2024, the reexamination of half of the cohort from SCAPIS1 started (the SCAPIS2). In SCAPIS2-HOME (a sub-study of SCAPIS2), individual responses to standardized isocaloric breakfasts and repeated Mixed Meal Tolerance Tests (MMTTs) will be investigated.

For this purpose, participants from the SCAPIS baseline cohort will be invited to take part in a 10-day intervention study, where participants will consume breakfast meals at clinic and the MMTTs at home. The breakfast meals will include ordinary cereal products that consist of either whole grain or refined grain foods served along with other typical breakfast items to be part of either a low-carbohydrate/high-fat or high-carbohydrate/low-fat breakfast. For the MMTTs, we will use standardized meal formulas called PhenFlex, which are high in calories, fat, and glucose and will be consumed repeatedly at home in the evening or the morning. Blood samples will be analyzed using clinical markers such as C-peptide, triglycerides, and markers of inflammation along with metabolomics. Continuous glucose monitoring will be used to obtain 24-hour interstitial glucose concentrations every 15 minutes during the 10-day intervention. Fecal- and blood samples will also be collected along with dietary assessments.

The research aims to understand the differential metabolic responses (glycemia, insulinemia, lipid profile, inflammation markers, and key metabolites) individuals may show after consuming whole grains or refined grains as part of breakfasts with high or low carbohydrate content. It is further to characterize to what extent an individual's specific characteristics, including the microbiota, health status, anthropometry, and habitual diet, drive such response differences. Since the study is a sub-set of the SCAPIS cohort, there are unique possibilities to relate the postprandial responses to hard risk factors such as prediabetic status (measured by oral glucose tolerance test), hepatic steatosis (liver fat deposition) and atherosclerotic plaque in the coronary arteries.

DETAILED DESCRIPTION:
The Swedish CArdioPulomonary bioImage Study (SCAPIS) is a national population study in Sweden, where comprehensive examinations have been carried out on 30,000 randomly selected people between 50-64 years during the years 2013-2018. The study is a collaboration between the country's six hospitals in Gothenburg, Malmö/Lund, Stockholm, Uppsala, Linköping and Umeå. The overall aim of SCAPIS is to reduce the risk of cardiovascular and pulmonary diseases in future generations. The study has resulted in a project where common diseases such as cardiovascular disease and chronic obstructive pulmonary disease (COPD) can be studied. SCAPIS research will better understand disease mechanisms and improve prevention and treatment methods.

SCAPIS 2 is a follow-up study conducted according to a detailed study protocol. Randomly selected participants from the SCAPIS baseline survey, 50% per site, will be invited to a re-survey until the desired number of 15,000 research subjects is reached. All research subjects will receive information about the study and informed consent will be obtained. The SCAPIS2-HOME study, will take place at two of the sites: Gothenburg and Umeå. In Gothenburg, 3133 participants will be examined over a two-year period, starting in January 2024. In Umeå, 1254 participants will be examined over the course of one year, starting in April 2024.

In SCAPIS2-HOME, all 4387 participants will go though a 10-day intervention where they will be provided with one standardized breakfast meal at the clinic and three mixed meal test drinks at home. The project will also include the collection of blood samples before and after meals to evaluate triglycerides, c-peptides, inflammation biomarkers (Glyc-A and hsCRP) along with metabolomics, continuous glucose monitoring, fecal samples and assessment of dietary intake.

During the first day of the intervention, the participants will be assigned to one of the four standardized meals. In Gothenburg, all standardised meals will be served in the morning, while in Umeå, half of the participants will consume the breakfast meals "as lunch". The meals will be based on foods regularly eaten for breakfast in Sweden, representing different carbohydrate and fat contents and containing either whole grain or refined grain products. One high fat/low carb (HF/LC) and one low fat/high carb (HF/LC) breakfast will be developed. The plan is to test different carbohydrate quality (whole grain vs. refined grain) for the HF/LC and the LF/HC breakfasts - resulting in four different breakfast meals.

In addition to the standardized breakfast meals, the participants will be instructed to perform three repeated Mixed Meal Tolerance Tests (MMTTs) at home. The PhenFlex drink will be used as MMTT in SCAPIS2-HOME which has been chosen to ensure our trial will be comparable with other large-scale trials planned in Europe currently. PhenFlex is a high-caloric mixed-meal challenge test containing 75 g of glucose, 60 g of fat, and 20 g of protein that induces a subtle systemic metabolic response.

The first MMTT should be done the day after the first clinical visit (Day 2), the second MMTT will take place three days after that (Day 5), and the third MMTT three days after that (Day 8). The participants will be randomized into two consumption patterns for the three MMTTs: morning, morning, evening (group 1), or evening, evening, morning (group 2). The randomization into the two groups for the MMTT tests are independent of which breakfast the participants has consumed.

Venous blood samples will be collected on the day at the clinic (Day 1). Capillary blood will be collected at the clinic and at home using collection kits from Capitainer® before and after the consumption of the standardized meal and the three meal tolerance tests. The samples will be collected at time 0, 60, 120 and 240 minutes.

A CGM (Abbott FreeStyle Libre Pro iQ [Chicago, Illinois, USA]) will be used to obtain Continuous glucose monitoring will be used to obtain 24-hour interstitial glucose concentrations every 15 minutes during the 10-day intervention.

Dietary intake will be assessed with a food frequency questionnaire previously used in SCAPIS (mini-MealQ) and with a repeated, web-based 24-hour recall (Riksmaten Flex from the Swedish Food Agency). The 24-hour recall will be filled in during the same four days as the test meals.

Lipemic and C-peptide responses (as a surrogate for insulin) will be measured in blood collected with Capitainers® before and after the meal challenge tests. Triglycerides will be measured with HPLC after lipid extraction. HDL, LDL, and other blood lipids will also be measured.

ELIGIBILITY:
Inclusion Criteria:

- Participants from the Swedish CArdioPulomonary bioImage Study (SCAPIS)

Exclusion Criteria:

* Food allergies or intolerances preventing consumption of any products included in the study
* Bariatric surgery, gastric bypass, or sleeve.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4387 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Continuous glucose monitoring (breakfast) | During breakfast day 1
  Differences in 24-hour CGM-measures and in the dynamic features of the postprandial glucose response as evaluated by CGM-home sampling between the different breakfasts
Lipemic responses (breakfast) | During breakfast day 1 (240 minutes)
  Differences in lipemic responses (triglycerides) as evaluated by home sampling between the different breakfasts
C-peptide (breakfast) | During breakfast day 1 (240 minutes)
  Differences in C-peptide responses as evaluated by home sampling between the different breakfasts
Glucose (breakfast) | During breakfast day 1 (240 minutes)
  Differences in glucose responses as evaluated by home sampling between the different breakfasts

SECONDARY OUTCOMES:
Inflammation markers (breakfast) | During breakfast day 1 (240 minutes)
  Differences in inflammation marker Glyc-A evaluated by home sampling between the different breakfasts
Inflammation marker (breakfast) | During breakfast day 1 (240 minutes)
  Differences in inflammation marker hsCRP as evaluated by home sampling between the different breakfasts
Continuous glucose monitoring (MMTT) | During intervention (day 2-8)
  Differences in 24-hour CGM-measures and in the dynamic features of the postprandial glucose response as evaluated by CGM-home sampling between morning and evening consumption of the mixed meal tolerance tests
Lipemic responses (MMTT) | During intervention (day 2-8)
  Differences in lipemic responses (triglycerides) as evaluated by home sampling between morning and evening consumption of the MMTTs
C-peptide (MMTT) | During intervention (day 2-8)
  Differences in C-peptide responses as evaluated by home sampling between between morning and evening consumption of the MMTTs
Glucose responses (MMTT) | During intervention (day 2-8)
  Differences in glucose responses as evaluated by home sampling between morning and evening consumption of the MMTTs
Inflammation markers (MMTT) | During intervention (day 2-8)
  Differences in inflammation markers (Glyc-A and hsCRP) as evaluated by home sampling between morning and evening consumption of the MMTTs
Continuous glucose monitoring (MMTT - interindividual) | During intervention (day 2-8)
  Interindividual differences in 24-hour CGM-measures and in the dynamic features of the postprandial glucose response as evaluated by CGM-home sampling between MMTTs consumed on the same timepoint (morning or evening) on different days
Lipemic responses (MMTT - interindividual) | During intervention (day 2-8)
  Differences in lipemic responses (triglycerides) as evaluated by home sampling between MMTTs consumed on the same timepoint (morning or evening) on different days
C-peptide (MMTT - interindividual) | During intervention (day 2-8)
  Differences in C-peptide responses as evaluated by home sampling between between MMTTs consumed on the same timepoint (morning or evening) on different days
Glucose (MMTT - interindividual) | During intervention (day 2-8)
  Differences in glucose responses as evaluated by home sampling between between MMTTs consumed on the same timepoint (morning or evening) on different days
Inflammation markers (MMTT - interindividual) | During intervention (day 2-8)
  Differences in inflammation markers (Glyc-A and hsCRP) as evaluated by home sampling between MMTTs consumed on the same timepoint (morning or evening) on different days
Correlation metabolic responses and microbiota | During the intervention (10 days)
  Correlations between metabolic responses (such as blood glucose, c-peptide, triglycerides, Glyc-A and CRP) from standardized meals with microbiota
Correlation metabolic responses and dietary intake | During the intervention (10 days)
  Correlations between metabolic responses (such as blood glucose, c-peptide, triglycerides, Glyc-A and CRP) from standardized meals and dietary intake measured from 24-hr recalls
Correlations metabolic responses and metabolome | During the intervention (10 days)
  Correlations between metabolic responses (such as blood glucose, c-peptide, triglycerides, Glyc-A and CRP) from standardized meals and the metabolome measured using metabolomics
Correlations metabolic responses and glucose tolerance | During the intervention (10 days)
  Correlations between metabolic responses (such as blood glucose, c-peptide, triglycerides, Glyc-A and CRP) from standardized meals and glucose tolerance measured using oral glucose tolerance test (OGTT)
Correlations metabolic responses and liver fat | During the intervention (10 days)
  Correlations between metabolic responses (such as blood glucose, c-peptide, triglycerides, Glyc-A and CRP) from standardized meals and liver fat
Correlations metabolic responses and atherosclerotic plaque | During the intervention (10 days)
  Correlations between metabolic responses (such as blood glucose, c-peptide, triglycerides, Glyc-A and CRP) from standardized meals and disease risk factors atherosclerotic plaque
Correlations metabolic responses and glucose | During the intervention (10 days)
  Correlations between metabolic responses (such as blood glucose, c-peptide, triglycerides, Glyc-A and CRP) from standardized meals and fasting blood glucose
Correlations metabolic responses and lipid status | During the intervention (10 days)
  Correlations between metabolic responses (such as blood glucose, c-peptide, triglycerides, Glyc-A and CRP) from standardized meals and fasting blood lipid status

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Region Västerbotten (Kliniskt Forskningscentrum), Umeå, Västerbotten County
  - Sahlgrenska University Hospital (Östra Hospital), Gothenburg, Västra Götaland County

IPD SHARING:
Plan to Share IPD: Undecided